CLINICAL TRIAL: NCT04987905
Title: The Effect of MIND-BE Program Applied to Intensive Care Nurses on Mental Health Parameters (Mindfulness Based Empowerment)
Brief Title: The Effect of MIND-BE Program on Mental Health Parameters (Mindfulness Based Empowerment)
Acronym: MIND-BE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Altundal (Other)
Collaborators: Mersin University (Other)
Responsible Party: Sponsor-Investigator, Hilal Altundal, Research Assistant, Principal Investigator, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hilal Altundal
Record Dates: First submitted 2021-07-28; First posted 2021-08-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Resilience; Posttraumatic Growth; Mindfulness; Self-compassion; Mental Health
Keywords: Resilience; Posttraumatic Growth; Mindfulness; Self-compassion; Mental health
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Participants and the researcher who carried out the application Hilal Altundal (H. A.) cannot be blinded due to the nature of the study. When the study is completed, the control and experimental groups will be coded as A and B and the data will be transferred to the computer environment by an independent researcher. The data coded as A and B will be analyzed by a statistician and the findings will be reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In the study, for 60 minutes once a week for 8 weeks the MIND-BE program will be applied to nurses. The program includes formal and informal practices of mindfulness ("Getting started, Introduction to MIND-BE, Noticing the autopilot, Power of attention, Simple awareness, Eating awareness, Body awareness, Breath awareness, Sitting awareness, Stress and reactions, Vision awareness, Challenging emotions and situations in business life, Awareness in business life, Awareness and communication, Awareness and compassion, Developing your own practice). In addition to these, nurses will be required to keep a diary of the program. This app contains basic mindfulness exercises and does not pose any health risks to practitioners. While the MIND-BE program is carried out in the online environment, the cameras of the nurses in the experimental group will be turned on and the researcher who made the application will be able to see each nurse.
  Interventions: Other: Mindfulness
- Control Group (No Intervention): No intervention will be made to the control group, only the data will be collected at the same time as the study group. After all data are collected (after the 12th week), the training content will be explained to the nurses in the control group and the MIND-BE program will be started for them as well. In this way, both groups will benefit from this program.

INTERVENTIONS:
Other: Mindfulness — In the study, for 60 minutes once a week for 8 weeks MIND-BE program will be applied to nurses. The program includes formal and informal practices of mindfulness ("Getting started, Introduction to MIND-BE, Noticing the autopilot, Power of attention, Simple awareness, Eating awareness, Body awareness, Breath awareness, Sitting awareness, Stress and reactions, Vision awareness, Challenging emotions and situations in business life, Awareness in business life, Awareness and communication, Awareness and compassion, Developing your own practice).
  Arms: Experimental Group

SUMMARY:
This study will be carried out in a pre-test-post-test, randomized controlled (parallel), experimental order in order to examine the effect of the MIND-BE program applied to intensive care nurses on mental health parameters. The hypothesis of this study is that MIND-BE program increases resilience, posttraumatic growth, mindfulness, self-compassion levels, and reduces mental symptoms.

DETAILED DESCRIPTION:
In the study, the MIND-BE program will be applied to the nurses (n=49) in the intervention group. Considering the studies on mindfulness on nurses, it is planned to practice mindfulness for 60 minutes once a week for 8 weeks. Mindfulness practice will be done online using appropriate platforms on the days and hours determined by Hilal Altundal (H.A.), who has a Mindfulness Institute-approved document. In the control group (n=49), no intervention will be made for 8 weeks. Results will be collected through data collection forms before the MIND-BE program, after the MIND-BE program is completed (8th week), and one month after the MIND-BE program is completed (12th week). The data collection forms applied to all nurses in the intervention and control groups at the beginning of the study will be applied again at the end of the 8th and 12th weeks. The primary expected outcome of the study is the effect of the MIND-BE program on nurses' resilience, posttraumatic growth, mindfulness, and self-compassion. The secondary expected result of the study is to determine the effect of the MIND-BE program on the mental health of nurses.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Written consent was obtained before participating in the study.
* Working as a nurse in the relevant institution on the dates of the study
* Not receiving any other psychological therapy during their working dates
* No prior meditation experience
* No practice in daily mind-body practices
* The participants (nurses) do not have any physical/mental disability or limitation and disease that would prevent them from participating in the program (no psychiatric diagnosis, no psychiatric medication, previous ear, brain, spinal cord surgery, acute retinal hemorrhage, vertebral fracture, and diaphragm rupture, hiatus or abdominal hernia, acute myocardial infarction, stable uncontrolled angina pectoris, severe coronary artery disease, congestive heart failure, severe valvular heart disease, acute myocarditis, acute and unstable musculoskeletal injuries, uncontrollable systemic hypertension, severe dementia and behavioral disorders) individuals are included in the study. will be included.

Exclusion Criteria:

* The participants (nurses) who could not complete eight sessions for different reasons and had to leave halfway through (illness, moving, changing service, etc.)
* The participants who participated in more than 70% of a mindfulness-based intervention prior to the study
* It is determined/specified that there are other existing health problems (physical/mental) after starting the education.
* Participating in less than 70% of the eight-week program
* Doing less than 70% of formal and informal practices
* Who left the program voluntarily

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Resilience will evaluate using The Resilience Scale for Adults | Change from before implementation, after mindfulness practice is completed (8th week), and one month after mindfulness practice is completed (12th week)
  It was developed by Friborg et al. The Turkish validity and reliability of the scale was done by Basım and Çetin. The 33-item scale consists of six sub-dimensions: "Self Perception", "Future Perception", "Structural Style", "Social Competence", "Family Cohesion" and "Social Resources". Opposite each item in the scale, there are five boxes with changing expressions for each question and showing a five-point Likert structure. Questions 1,3,4,8,11,12,13,14,15,16,23,24,25,27,31,33 in the scale without any cutoff point are reverse coded. The scoring of the boxes ranges from 1 to 5 for flat coded items; from 5 to 1 for reverse coded items. The total Cronbach's alpha coefficient of the scale is 0.86, and the Cronbach's alpha coefficients of the sub-dimensions range from 0.66 to 0.81.
Posttraumatic growth will evaluate using The Post Traumatic Growth Inventory | Change from before implementation, after mindfulness practice is completed (8th week), and one month after mindfulness practice is completed (12th week)
  It was developed by Tedeschi and Calhoun (1996). The Turkish validity and reliability of the scale was done by Kağan et al. (2012). Consisting of 21 items in total, the scale has a six-grade Likert structure (No way (0), Very little (1), A little (2), Moderate (3), Quite a lot (4), Very much (5)) . The scale consists of three sub-dimensions: "self-perception", "change in philosophy of life" and "relationship with others". An increase in the scores obtained from the scale without any cut-off point indicates that the level of post-traumatic growth increases. Similarly, the increase in the scores obtained from the sub-dimensions indicates that the sub-dimensions with increasing scores are used more. The Cronbach's alpha values of the scale ranged from 0.92, and the Cronbach's alpha values of the sub-dimensions ranged from 0.77 to 0.88.
Mindfulness will evaluate using The Mindful Attention Awareness Scale | Change from before implementation, after mindfulness practice is completed (8th week), and one month after mindfulness practice is completed (12th week)
  The Mindful Attention Awareness Scale (MAAS), developed by Brown and Ryan (2003), is a 15-item scale that measures the general tendency to be aware of and attentive to momentary experiences in daily life. MAAS has a single factor structure and gives a single total score. High scores on the scale indicate high conscious awareness. The MAAS is a 6-point Likert-type scale (almost always, often, sometimes, rarely, quite rarely, almost never). The internal consistency coefficient was determined as 0.80 in the Turkish adaptation study of the MAAS by Özçiçek et al. (2011).
Self-compassion will evaluate using The self-compassion scale | Change from before implementation, after mindfulness practice is completed (8th week), and one month after mindfulness practice is completed (12th week)
  Developed by Neff (2003), Akın et al. (2007), the self-compassion scale (self-compassion scale) consists of 26 items and six subscales (self-compassion, self-judgment, shared human experience, isolation, mindfulness, and hyper-identification). In this scale, which has a five-point Likert-type rating; almost never (1), rarely, sometimes, often, almost always (5). In the study of Akın et al. (2007), the internal consistency of the subscales ranged between 0.72 and 0.80.

SECONDARY OUTCOMES:
Mental symptom will evaluate using The Brief Symptom Inventory | Change from before implementation, after mindfulness practice is completed (8th week), and one month after mindfulness practice is completed (12th week)
  The Brief Symptom Inventory (BSI) is based on the 90-item Symptom Check List (SCL-90) distributed over nine factors, and is a 53-item scale consisting of the items with the highest load in each factor. The scale is a Likert-type self-evaluation inventory developed by Deregotis in 1992. The scale is the short form of the Mental Symptom Checklist and consists of five subscales and three global indexes. As a result of these studies, in the Turkish adaptation of the scale by Şahin and Durak (2002), the BSI was organized into five subsections as "Anxiety", "Depression", "Negative Self", "Somatization" and "Hostility". An increase in the total score indicates an increase in the weight of the question. There is no cut-off value for BSI. The alpha coefficients found for the subscales of BSI in the study were Depression, α=0.88; anxiety, α=0.87; negative self, α=0.87; somatization, α=0.75; hostility is listed as α=0.76. The points that can be obtained from the inventory range from 0 to 212.

CONTACTS AND LOCATIONS:
Overall Officials: Mualla Yılmaz, Professor, Study Director — Mersin University, Faculty of Nursing, Ciftlikkoy Campus, 33343, Yenisehir, Mersin
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No